CLINICAL TRIAL: NCT05017428
Title: Absorption and Digestion Kinetics of Human Metabolites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Angela Zivkovic, PhD, Associate Professor, University of California, Davis
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1725738
Record Dates: First submitted 2021-08-11; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Postprandial Inflammation
MeSH Terms: interventions — Spermidine; Niacinamide; Flour

STUDY DESIGN:
Intervention Model Description: Participants will take a supplement containing 4 metabolites at escalating doses compared with placebo after a standardized meal and their blood will be drawn at mutliple points throughout a postprandial time course to evaluate markers of inflammation, circulating levels of each metabolite, and plasma functionalities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose (Experimental): The Low Dose arm provides subjects with supplementation with 5mg of spermidine (in the form of 5g of a 0.1% spermidine wheat germ extract), 500mg of nicotinamide, 400mg of palmitoylethanolamide, and 200mg of oleoylethanolamide.
  Interventions: Dietary Supplement: Spermidine; Dietary Supplement: Nicotinamide; Dietary Supplement: PEA; Dietary Supplement: OEA
- Medium Dose (Experimental): The Medium Dose arm provides subjects with supplementation with 10mg of spermidine (in the form of 10g of a 0.1% spermidine wheat germ extract), 750mg of nicotinamide, 800mg of palmitoylethanolamide, and 400mg of oleoylethanolamide.
  Interventions: Dietary Supplement: Spermidine; Dietary Supplement: Nicotinamide; Dietary Supplement: PEA; Dietary Supplement: OEA
- High Dose (Experimental): The Low Dose arm provides subjects with supplementation with 15mg of spermidine (in the form of 15g of a 0.1% spermidine wheat germ extract), 1000mg of nicotinamide, 1200mg of palmitoylethanolamide, and 600mg of oleoylethanolamide.
  Interventions: Dietary Supplement: Spermidine; Dietary Supplement: Nicotinamide; Dietary Supplement: PEA; Dietary Supplement: OEA
- Placebo (Placebo Comparator): In this arm the participants are given supplementation with a placebo control consisting of 15g of wheat flour.
  Interventions: Dietary Supplement: Wheat Flour

INTERVENTIONS:
Dietary Supplement: Spermidine — Spermidine in the form of a 0.1% spermidine wheat germ extract
  Other Names: Primeadine
  Arms: High Dose; Low Dose; Medium Dose
Dietary Supplement: Nicotinamide — Nicotinamide given as niacinamide
  Other Names: Jarrow Niacinamide
  Arms: High Dose; Low Dose; Medium Dose
Dietary Supplement: PEA — Palmitoylethanolamide given at 98% purity
  Other Names: Nootropics Depot PEA
  Arms: High Dose; Low Dose; Medium Dose
Dietary Supplement: OEA — Oleoylehtanolamide given at 90% purity
  Other Names: Riduzone
  Arms: High Dose; Low Dose; Medium Dose
Dietary Supplement: Wheat Flour — Wheat flour given as a placebo control
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to evaluate the effects oral supplementation with four human metabolites (spermidine, nicotinamide, palmitoylethanolamide (PEA), and oleoylethanolamide(OEA)) at varying doses on the circulating blood levels of these metabolites as well as their immediate effects on plasma functionality and postprandial inflammation. 5 young healthy subjects will participate in a four armed study consisting of a Placebo arm and a Low, Medium, and High Dose arm. Subjects will be given a standardized breakfast along with supplementation with either an escalating dose (Low: 1x, Medium: 2x, High: 3x) of a combination of spermidine, nicotinamide, PEA and OEA or a placebo control and a time course of their blood plasma will be collected after supplementation. Plasma samples will be assessed for their concentration of spermidine, nicotinamide, PEA, and OEA as well as their experimental and clinical functionalities including their anti-inflammatory, antioxidant, and cholesterol efflux abilities on primary human macrophage.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 years old to constitute a young study population
* BMI: 19-27 kg/m2 to constitute a normal/healthy weight population
* Weight: 133lbs or more
* Subjects must be willing and able to consume a standardized breakfast bar containing cashews and dates (Larabar).
* Subjects must be willing to consume oral dietary supplement versions of spermidine, 1-methlynicotinamide, palmitoylethanolamide, and oleoylethanolamide.
* Subjects must be willing and able to undergo blood draws at the UC Davis Ragle Nutrition Center at 0, 1, 2, and 4 hours after supplementation with spermidine, niacinamide, palmitoylethanolamide, and oleoylethanolamide.

Exclusion Criteria:

* Smoker
* Anemia
* Documented chronic diseases including diabetes, thyroid disease, metabolic syndrome, cancer, autoimmune diseases, or previous cardiovascular events
* Any inflammatory bowel disease including IBS, Crohn's Disease, Celiac Disease
* Any allergy or sensitivity to wheat, gluten, or soy products
* Consumption of >1 alcoholic drink/day
* Current consumption of any probiotic, prebiotic, or dietary supplements
* Extreme dietary or exercise patterns
* Recent weight fluctuations (greater than 10% in the last six months)
* Regular use of over-the-counter allergy or pain medications (>1/week)
* Taking prescription lipid medications (e.g. statins) or other supplements known to alter lipoprotein metabolism such as isoflavones.
* Use of any form of hormonal birth control including oral contraception pills, hormonal IUDs or rings, or hormonal birth control patches
* Illness such as flu or cold of any kind within the last two weeks
* Allergy to components of standardized breakfast bar (cashew/dates)
* Changes to any of the above during the study period.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participation in the study will be restricted to males. Women will be excluded from the study as the study protocol includes multiple study arms to be completed within a 1 month timeframe. Biological variations caused by the menstrual cycle throughout a single month may cause week to week variability in the absorption, digestion, and metabolism of our metabolites of interest that cannot be controlled for in this small pilot study.
Enrollment: 5 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Circulating Plasma Levels of Metabolites | 1, 2, and 4 hours after ingestion
  Quantitative plasma concentrations of spermidine, nicotinamide, pamitoylethanolamide, and oleoylethanolamide (in nmol/L).

SECONDARY OUTCOMES:
Anti-inflammatory capacity of plasma | 1, 2, and 4 hours after ingestion
  Ex vivo assessment of the effects of subject plasma on the secretion of pro-inflammatory cytokine TNF-alpha (pg/mL) by primary human macrophage

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rhodes CH, Hong BV, Tang X, Weng CY, Kang JW, Agus JK, Lebrilla CB, Zivkovic AM. Absorption, anti-inflammatory, antioxidant, and cardioprotective impacts of a novel fasting mimetic containing spermidine, nicotinamide, palmitoylethanolamide, and oleoylethanolamide: A pilot dose-escalation study in healthy young adult men. Nutr Res. 2024 Dec;132:125-135. doi: 10.1016/j.nutres.2024.10.006. Epub 2024 Oct 23. PMID 39549554